CLINICAL TRIAL: NCT05945979
Title: Avaliação da eficácia de um Novo Suplemento Alimentar Para Cabelos e Unhas- Estudo in Vitro, clínico, Subjetivo e Instrumental
Brief Title: Evaluation of the Efficacy of a New Supplement for Hair and Nails - in Vitro, Clinical, Subjective and Instrumental Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Farmoquimica S.A. (Industry)
Collaborators: Kosmoscience Ciência e Tecnologia Cosmética Ltda (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FQM166-20
Record Dates: First submitted 2023-05-26; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-06

CONDITIONS: Hair Loss; Nails, Ingrown
Keywords: capillary density; strengthening; hair loss
MeSH Terms: conditions — Alopecia; Nails, Ingrown | interventions — Biotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A power supplement with biotin (Experimental): 40 participants using the product for 90 days. Aims to evaluate the clinical, subjective and instrumental usage
  Interventions: Dietary Supplement: A power supplement with biotin

INTERVENTIONS:
Dietary Supplement: A power supplement with biotin — A power dietary supplement containing aminoacids and vitamins

SUMMARY:
A unicentric, exploratory, prospective clinical an in vitro study to evaluate efficacy and safety of a Supplement in improving the quality and general aspects of hair and nails in female participants through clinical,in vitro, subjective and instrumental evaluations

DETAILED DESCRIPTION:
A unicentric, exploratory, prospective clinical an in vitro study to evaluate efficacy and safety of a Supplement in improving the quality and general aspects of hair and nails in female participants through clinical, in vitro, subjective and instrumental evaluations.

It will be necessary 40 female participants aged between 25 and 55 years old with a clinical and in vitro diagnosis of telogen effluvium presenting at least one of the following characteristics: hair loss problems caused by stress, poor diet and excess of tinctures and chemicals procedures applied to hair, and menopausal women.

The participants will remain in the study for 93 days using the product. Visits will be scheduled in D-3, D0, D45, D48, D90, D93.

Instrumental evaluations: Evaluated on each visit:

* To analyze the biological cycle of hair growth using Trichogram test - D-3, D45, D90;
* Evaluation of hair growth kinetics using phototrichogram - D-3,D0, D45, D48, D90, D93;
* Evaluation of the mechanical strength of the hair structure using EMIC DL 500- D-3, D90
* Evaluation of the dermal density of the scalp using the high-frequency ultrasound- D-3, D45, D90
* Participants will respond to a subjective assessment using a questionnaire to capture a subjective efficacy- D45, D90

ELIGIBILITY:
Inclusion Criteria:

* Phototype (Fitzpatrick): I to VI.
* Have intact skin in the test region: scalp.
* Present a clinical diagnosis of telogen effluvium.
* Agree to adhere to the study procedures and requirements: study time, returns (D-3, D0, D45, D48,D90 and D93) to the laboratory to carry out the study procedures, administration of the product research, fill the use diary, fill the perceived efficacy questionnaire, carrying out the collection of hair samples (hair cut, close to the scalp - beginning of the study and after 90 days), not change hair habits during the study period.
* Agree not to carry out chemical hair treatments (hair coloring, straightening, among others) and/or treatment to control/reduce hair loss and/or dandruff, among others, until the end of the study (90 days).
* Agree with the procedure for collecting hair samples: trichogram and hair cut, close to the leather hairy.
* Agree to administer 01 capsule/day of the investigational product. Present a minimum length of hair (3 cm) to carry out the procedure for collecting samples of hair
* Present hair and brittleness for at least 3 months before the start of the study.
* Signature of the Free and Informed Consent Term (TCLE).

Exclusion Criteria:

* Pregnancy
* During the course of the study, the subject develops symptoms of COVID-19, such as: fever (temperature above 37.5°C), cough; dyspnoea (difficulty breathing characterized by rapid, short breaths, usually associated with heart or lung disease); myalgia (muscle pain); upper respiratory symptoms; fatigue and more rarely, gastrointestinal symptoms.
* Appearance of disease that requires the use of medications prohibited in this protocol: use of corticoids and anti-inflammatories for a period longer than 15 days and/or in high doses (above 1mg/kg).
* Use of immunosuppressants during the study period.
* Use of Vitamin A or its derivatives and other vitamins and minerals.
* Beginning or changing hormone treatments after signing the TCLE.
* Swallowing difficulty: dysphagia.
* Presence of dermatoses or active skin lesions (local and/or disseminated) in the study region.
* Hypersensitivity reactions (allergic reactions, irritation or feelings of discomfort) caused by actives or excipients from the investigational product.
* Vaccine use during the study period.
* Diagnosis of diabetes or nephropathies during the study period.

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Evaluate efficacy of a power supplement in reducing hair loss throgh thichogram analysis | Day 93
  Evaluate the effectiveness of the product investigational in providing reduction of hair loss through thrichogram analysis. If the ratio between anagen/telogen hairs strands is > 4, it indicates improvement in reducing hair loss after daily and continuous use for a period of up to 90 days.

SECONDARY OUTCOMES:
Analysis of the biological cycle of hair growth- Trichogram | Three days before the beginning of product intake, Day 45 and Day 90
  Evaluate the phase of the biological cycle of hair growth (anagen, telogen or catagen) and determine the ratio between anagen/telogen hair strands. If the ratio between anagen/telogen hairs strands is ≤ 4, it indicates positive symptoms for androgenetic alopecia or telogen effluvium and the partipant will be included in the study.The trichogram was performed three days before the beginning of product intake, and after 45 days and 90 days of continuous use.
Evaluation of hair growth kinetics- Phototrichogram | Three days before the beginning of product intake, Day 0, Day 45, Day 48, Day 90 and Day 93
  Evaluate the growth kinetics of hair strands after shaving a standardized area of 1 cm² of the scalp and taking images on the same day and three days after. In total, three scrapings were performed on three days before intervention, day 45 and day 90, totaling six image collections. A microscope (i-Scope USB, Moritex, JP) with a 30x lens and polarized light was used to obtain the images. In each collection, three microimages of the evaluated area on the head of each participant were recorded.
Monitoring of hair growth by photographic documentation | Day 0, Day 45 and Day 90
  Evaluation of the dermal thickness of hair strands through specific software. Patients will be submitted to the Ultrascan UC 22 MHz equipment (Courage + Khazaka electronic GmbH), on day 0 and after 45 days and 90 days of continuous use of the investigational product.
Evaluation of the mechanical strength of the hair structure using EMIC DL 500 | Three days before the beginning of product intake and Day 90
  Evaluation of the mechanical resistance of the hair. 50 hairs strands were collected from each participant and cut with the aid of scissors to avoid possible damage to the hair shaft resulting from traction for pulling out. The test was performed three days before the beginning of product intake and after 90 days of continuous use.
Subjective efficacy of the participants by questionnaire | Day 45 and Day 90
  Evaluate the perceived efficacy of the product from the participant's point of view through a subjective questionnaire after 45 days e 90 days of continuous use of the product. The questionnaire uses a 7-point scale, where 1 meaning poor and 7 means excellent.

CONTACTS AND LOCATIONS:
Locations (1):
- Kosmoscience Ciência e Tecnologia Cosmética Ltda, Valinhos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: D93